CLINICAL TRIAL: NCT05183711
Title: Self-Evaluating Anesthesia Competency Among Nurse Anesthetists: The Survey Study
Brief Title: Self-Evaluating Anesthesia Competency Among Nurse Anesthetists
Status: Completed | Type: Observational
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Ngamjit Pattaravit, ASST. PROF, Prince of Songkla University
Other Study IDs: competency self evaluation
Record Dates: First submitted 2020-01-31; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Anesthesia Competences (Self-evaluation)
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Nurse anesthetist: In this study, the investigator team designs to use self-evaluating form as a tool for any competencies evaluation. The Numerical Rating Scale (range from 1-10, 1= least competency, 10 =highest competency) will be used for any anesthesia skills evaluation. The participant could download the self-evaluating form (google form, no personal identity record) via QR code.
  Interventions: Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: Questionnaires — The Numerical Rating Scale (range from 1-10, 1= least competency, 10 =highest competency) will be used for any anesthesia skills evaluation. (download the self-evaluating form via QR code)

SUMMARY:
Continuing Medical Education (CME) has been proved that not only improving healthcare provider performance but also improving the patient outcome.Previous studies results showed that long established and multiple CME sessions, various methods and interactive sessions help the learners to improve their competency. CME among the nurses seem to be more difficult than in the physicians. Regarding to work schedule, lack of support from institution especially funding. Outcome-based continuing professional development course that provide practical skills sessions and give a chance for learners to reflect themselves help the learner to determine the performance gap between the learner real life practice and the standard of care. So in term of professional development, the practitioner can improve their competency from clinical level to professional level and finally managerial level.

After graduation,There are just only few anesthesia education courses for nurse anesthetists in each year. These may be not enough in order to maintain either knowledge or essential skills needed in anesthesia real life practice. The primary objective of this is to determine that which kinds of knowledge and skills in anesthesia that the nurse anesthetists in our institution lack off.

DETAILED DESCRIPTION:
After graduation, CME is one of the important step to improve both the graduate's competencies and the quality of healthcare services. Throughout the professional career paths, nurse anesthetists in different career stages have different level of competency and expectations. Retention of knowledge and skills are much different between the new graduate nurses and mid to late career nurse. Feasible training program by using interactive teaching methods can improve the learner's satisfaction. There are just only few anesthesia education courses for nurse anesthetists in each year. These may be not enough in order to maintain either knowledge or essential skills needed in anesthesia real life practice. The primary objective of this is to determine that which kinds of knowledge and skills in anesthesia that the nurse anesthetists in our institution lack off. The secondary objective is the correlation between anesthesia non-technical skills (ANTS) and years of experience among nurse anesthetists. The results of this study will be useful information for creating additional anesthesia training course for this graduate group. Furthermore, Improving the anesthesia standard of care in the near future.

In this study, the investigator team designs to use self-evaluating form as a tool for any competencies evaluation. The Numerical Rating Scale (range from 1-10, 1= least competency, 10 =highest competency) will be used. After ethical committee approval, the subject group will be invited by the investigator team by using participant information form. In case of the participants have willing to enroll in this study. The consent form must be signed and then the participant could download the self-evaluating form (google form, no personal identity record) via QR code. After data collection completion, the statistical analysis will be done by using R program. The statistically significance is set as p< 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Nurse anesthetist at Prince of Songkla Hospital who is currently working in Anesthesia field

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: -Nurse anesthetist at Prince of Songkla Hospital who is currently working in Anesthesia field
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2019-11-25 (Actual)

PRIMARY OUTCOMES:
determine level of knowledge and skills in anesthesia among nurse anesthetists | from 0 to 35 years of experience in anesthesia
  level of competency (1-10)

SECONDARY OUTCOMES:
correlation between anesthesia non-technical skills (ANTS) and years of experience among nurse anesthetists. | from 0 to 35 years of experience in anesthesia
  correlation between anesthesia non-technical skills (ANTS) and years of experience among nurse anesthetists.

CONTACTS AND LOCATIONS:
Overall Officials: ngamjit pattaravit, MD, Principal Investigator — Prince of Songkla University
Locations (1):
- Prince of Songkla University, Hat Yai, Changwat Songkhla, Thailand

IPD SHARING:
Plan to Share IPD: No